CLINICAL TRIAL: NCT06037720
Title: Diagnostic Accuracy Study of a Point-of-Care Test for Coagulation Function: CoaguChek System Versus Standard Laboratory Tests in Cardiac Surgery Requiring Cardiopulmonary Bypass
Brief Title: Diagnostic Accuracy Study of a Point-of-Care Test for Coagulation Function
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, Fabricio Tavares Mendonca, MD, MSc, PhD, Hospital de Base
Other Study IDs: PeriopCoaguChek
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: CoaguChek® XS System; Coagulation Function
Keywords: CoaguChek® XS System; International normalized ratio; Point-of-care testing; Cardiopulmonary bypass

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Coaguchek testing — Patients scheduled electively to undergo cardiac surgery with cardiopulmonary bypass at Hospital de Base in the Federal District.

SUMMARY:
Intraoperative coagulopathies in complex procedures are common. For the diagnosis and adequate therapy, laboratory tests are necessary, which can delay the patient's therapy. In this sense, the study aims to evaluate the point-of-care test device for patients undergoing surgeries with cardiopulmonary bypass.

Objective: To analyze the accuracy between the point-of-care diagnostic method and the laboratory test considered the gold standard for checking the INR.

Methodology: Cross-sectional study of diagnostic accuracy with simultaneous testing of the Coaguchek XS device and standard laboratory method in patients undergoing cardiopulmonary bypass to evaluate INR results.

DETAILED DESCRIPTION:
Laboratory evaluation of blood clotting is widely used in perioperative medicine, either by conventional technique (prothrombin time - PT/INR, Activated Partial Thromboplastin Time - aPTT, fibrinogen dosage and platelet count) or by the Point of Care method (Thromboelastogram ) - notably in surgical procedures with the possibility of severe volume loss (cardiovascular, oncological, trauma, etc.).

The prothrombin time (PT) is a general assessment of the integrity of the extrinsic and common pathway of coagulation. It determines the time of formation of the fibrin clot. The INR/RNI (International Normalized Ratio) is calculated from the PT and is intended to establish valid comparisons regardless of the type of PT reagent (known as thromboplastin) used by different clinical laboratories. The INR is indicated for evaluating the integrity of the extrinsic (factor VII*) and common pathway (fibrinogen and factors II*, V and X*), and for monitoring the anticoagulant effect of an anti-vitamin K agent (warfarin), capable of inhibiting the synthesis of vitamin K dependent factors (II, VII, IX, X, proteins C and S).

Today, due to its safety, sensitivity and speed, the thromboelastogram is recommended as the method of choice for assessing hemostasis in a surgical setting. However, because it is still not widespread in many centers, mainly due to its high cost, many hospitals are limited to the use of traditional laboratory methods which, despite their undeniable reliability, require more time for their execution and release of results.

In cardiac surgery with cardiopulmonary bypass (CPB), the use of prime solution to fill the CPB circuit results in hemodilution of coagulation factors, with factor I (fibrinogen) being one of the most affected, but not the only one. Each abnormality detected requires a specific action. Thus, the activated clotting time (ACT) is normalized with the administration of protamine. Thrombocytopenia and/or platelet dysfunction, with platelet concentrate infusion. Abnormalities in clotting factors, with administration of the specific factor, eg fibrinogen, either by factor concentrate, cryoprecipitate or plasma. It is at this moment that a quick assessment of hemostasis, in a global and individualized way at the same time, is necessary.

More than a decade ago, devices appeared on the market designed to help patients using warfarin to maintain their anticoagulation within parameters established for each case, providing safety, speed and comfort. Using a reagent strip and a drop of blood, evaluating the INR has become as simple as evaluating capillary blood glucose for diabetic patients. In just a few seconds, INR assessment can show significant changes in the extrinsic coagulation pathway, an important step to help with rapid decision-making in surgical environments. The Coaguchek Device, validated and used for outpatient management of patients using Warfarin, presents valuable characteristics for this purpose (simplicity, speed, safety), also important in the context of intraoperative decision-making. There are few reports in the literature on the use of the Coaguchek device in surgery and on the reliability of the data obtained through its use.

To evaluate this correlation, the main objective of the present study is to evaluate the effectiveness of the portable INR meter in a surgical setting and comparing it with conventional laboratory methods. The proposal is a cross-sectional diagnostic study in patients scheduled electively to undergo cardiac surgery with cardiopulmonary bypass at Hospital de Base in the Federal District.

All patients will receive standard monitoring associated with hemodynamic monitoring with invasive blood pressure and central venous access. Balanced general inhalation anesthesia will be administered to all patients. Hemodynamic support with dobutamine, noradrenaline, nitroprusside, nitroglycerin, vasopressin, or milrinone will be offered according to perioperative needs. The same commercial brand of heparin and protamine will be used to all the patients.

Laboratory tests, including samples for the Coaguchek device strip, will be collected 10 minutes before heparin administration and 10 minutes after the end of the protamine infusion. The laboratory exams that will be collected are: arterial blood gases, venous blood gases, electrolytes, complete blood count, coagulogram (TAP, aPTT, INR) and fibrinogen.

The sample size was calculated for the limits of agreement by Bland and Altman (1986)1, according to the method developed by Lu et al. (2016).2 Based on previous studies3-5, we assumed a mean difference between the POC test and the laboratory test of 0.126 units with a standard deviation of 0.132. Furthermore, based on clinical criteria, we consider that an absolute difference greater than 0.5 units will be clinically relevant. In other words, the maximum difference (Δ) between the tests (so as not to change the clinical approach) would be up to ± 0.5 units; that is, (-Δ ,Δ) equals (-0.5,0.5). Assuming a 5% ɑ level and 95% confidence intervals around the Bland-Altman limits of agreement, 43 participants were needed to ensure a statistical power of 90% to detect agreement between the two methods. All calculations were performed using the Stata 16 program (StataCorp, Texas, United States). We decided to increase the sample to 50 patients for cases of loss to follow-up or failures in annotations.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* admitted to the Hospital de Base of the Federal District for cardiac surgery, who volunteered to participate in the examination both by the traditional method of venous INR examination and by the use of the Coaguchek device and only after signing the TCLE.

Exclusion Criteria:

* patients who give up the research even after signing the TCLE will be excluded
* patients who do not meet the aforementioned inclusion criteria
* patients who refuse to participate in the study
* patients with kidney, liver, hematological disease or any disease that affects coagulation
* patients participating in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled electively to undergo cardiac surgery with cardiopulmonary bypass at Hospital de Base in the Federal District.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Point-of-care diagnostic method | During surgery
  To analyze the accuracy between the point-of-care diagnostic method and the laboratory test considered the gold standard for verifying the INR.

REFERENCES:
- [Background] Khalaf-Adeli E, Alavi M, Alizadeh-Ghavidel A, Pourfathollah AA. Comparison of standard coagulation testing with thromboelastometry tests in cardiac surgery. J Cardiovasc Thorac Res. 2019;11(4):300-304. doi: 10.15171/jcvtr.2019.48. Epub 2019 Oct 13. PMID 31824611
- [Derived] Mendonca FT, Matos SH, Moreira LG, Pereira IL, Dino LL, Braga MB, Dias GHDS. Accuracy of a point-of-care CoaguChek test versus standard laboratory coagulation monitoring in cardiac surgery involving cardiopulmonary bypass: randomized clinical trial. Braz J Anesthesiol. 2025 Nov 22;76(2):844714. doi: 10.1016/j.bjane.2025.844714. Online ahead of print. PMID 41276168